CLINICAL TRIAL: NCT02127463
Title: Phase II/III Study of the Efficacy and Safety of MacuCLEAR MC-1101 1.0% BID in the Treatment of Non-exudative Age-Related Macular Degeneration
Brief Title: Phase II/III Study of the Efficacy and Safety of MacuCLEAR MC-1101 in Treating DryAge-Related Macular Degeneration
Acronym: McCP2/3
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MacuCLEAR, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC-1101-003
Record Dates: First submitted 2014-04-25; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Non-Exudative Age Related Macular Degeneration
Keywords: AMD; Dry AMD; Non-Exudative AMD; MC-1101
MeSH Terms: interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MC-1101 active (Experimental): Topical Drug 1% Ophthalmic Solution Topically, two times per day; morning and bedtime
  Interventions: Drug: MC-1101
- MC-1101 Vehicle Control (Placebo Comparator): Topical Drug:
  Ophthalmic Solution Topically, two times per day; morning and bedtime
  Interventions: Drug: MC-1101 Vehicle

INTERVENTIONS:
Drug: MC-1101 — Topically, two times a day, morning and bedtime
  Other Names: 1% Ophthalmic Solution
  Arms: MC-1101 active
Drug: MC-1101 Vehicle — Topically, two times a day; morning and bedtime
  Other Names: Topical Ophthalmic Solution
  Arms: MC-1101 Vehicle Control

SUMMARY:
This is a Phase II/III,vehicle controlled, double masked, single center study. A single eye of 60 individuals with mild to moderate non-exudative Age-Related Macular Degeneration (AMD) will be randomly assigned to receive either topical 1% MC-1101 or a vehicle control over 2 years. The study design will assess the efficacy, safety, and tolerability of MC-1101 for these patients.

An analysis of the primary and secondary endpoints will be conducted when all subjects have completed Baseline, 1, 3, 6, 12,18 and 24 months.

DETAILED DESCRIPTION:
MC-1101is a topically administered drug which in previous clinical studies has been proven to get to the back of the eye. MC-1101is a 505 (b) 2 compound and has FDA Fast Track Status. It is a strong, vasoactive drug which is intended to increase choroidal blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age ≥ 50 years and ≤ 85 years
* Females only: At least 1year since last menstrual period or surgically sterilized
* 20/80 or better ETDRS best corrected visual acuity
* Early to intermediate nonexudative AMD (AMD category 3 through 3b on Age-Related Eye Disease Study (AREDS) Report No. 8 AMD Categories
* Willing and able to sign informed consent, comply with study protocol requirements, and undergo at least 2.5 hours of testing at each visit
* Able to reliably to complete biophysical testing
* Willing to take an AREDS2 based formula vitamin as indicated

Exclusion Criteria:

* Past or current exudative AMD or central geographic atrophy in study eye; (AMD Category 4 on Age-Related Eye Disease Study (AREDS) Report No. 8 AMD Categories)
* Past or current retinal or choroidal vasculopathy in study eye (e.g. serous or hemorrhagic pigment epithelial detachment, polypoidal choroidal vasculopathy, central serous chorioretinopathy, retinal vein occlusion, sickle cell retinopathy)
* Uncontrolled hypertension (≥ 160 systolic or ≥95 diastolic)
* Glaucoma
* Dilated pupil diameter less than 6 millimeters
* Subjects with a history of a hypersensitivity reaction to the study drug or to any agent used in the components of the study assessment
* Use of topical ocular medications (other than artificial tear products)
* Anticipated extra- or intraocular intervention during the study period
* High myopia (refractive error spherical equivalent ≥ -6 diopters)
* Optic neuropathy
* Neurological conditions that can impair vision (e.g. Parkinson's disease, multiple sclerosis, Alzheimer's disease)
* Liver disease (e.g. cirrhosis, hepatitis)
* History of small bowel surgery
* Current or past use for more than 30 days of chloroquine, hydroxychloroquine, chlorpromazine, thioridazine, quinine sulfate, clofazimine, cisplatin, carmustine (BCNU), deferoxamine, amiodorone, isoretinoin, or gold
* Contact lens wearers (not prepared to discontinue lens use)
* Ophthalmic surgery of any kind within 3 months prior to screening visit
* Participation in any interventional clinical study requiring IRB approval within 3 months prior to screening visit of this study
* Currently being treated for cancer or any disease likely to adversely affect participation in a 2 year study
* Known to have AIDS/HIV
* Current use of hydralazine
* Any other findings deemed unacceptable by the Principal Investigator or Sponsor

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Visual Function | Up to 24 months
  Primary efficacy assessment will be a comparison between groups of the change in visual function at 12 months with additional analyses at 18 and 24 months measured by dark adaptation methodology.

SECONDARY OUTCOMES:
Safety and tolerability (incidence and severity of adverse events, ocular irritability, ocular hyperemia) | Up to 24 months
  Evaluate the safety and tolerability (incidence and severity of adverse events, ocular irritability and ocular hyperemia) of MC-1101compared to a vehicle control at each study visit following treatment for 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell J Goff, MD, Principal Investigator — Rocky Mountain Retina Consultants
Locations (1):
- Rocky Mountain Retina Consultants, Murray, Utah, United States